CLINICAL TRIAL: NCT06894901
Title: Assessing the Efficacy of Incompatible Insect Technique Coupled with Sterile Insect Technique (IIT-SIT) to Manage Large Dengue Clusters: a Randomized Controlled Trial
Brief Title: Impact of IIT-SIT on Dengue Clusters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Environment Agency, Singapore (Other Government)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Lee Ching Ng, Group Director (Environmental Health Institute), National Environment Agency, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2025
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention clusters (Experimental): Dengue clusters in residential estates that receive releases of male Wolbachia-infected Aedes aegypti
  Interventions: Biological: Biological (Male Wolbachia-infected Aedes aegypti)
- Non-intervention clusters (No Intervention): Dengue clusters in residential estates that do not receive releases of male Wolbachia-infected Aedes aegypti

INTERVENTIONS:
Biological: Biological (Male Wolbachia-infected Aedes aegypti) — Releases of male Wolbachia-infected Aedes aegypti mosquitoes
  Arms: Intervention clusters

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of Wolbachia-infected male mosquitoes combined with sterile insect technique (IIT-SIT) to mitigate active dengue transmission in Singapore.

DETAILED DESCRIPTION:
Aedes-borne diseases are expected to increase in geographical coverage and intensity due to climate change and rapid urbanization. It has been demonstrated that Wolbachia-mediated incompatible insect technique coupled with sterile insect technique (IIT-SIT) is highly effective in suppressing Aedes populations and subsequently reducing dengue risk. However, the efficacy of the tool in mitigating ongoing transmission is unknown.

The researchers outline a randomized controlled trial to be conducted in high-rise public housing estates in Singapore to assess the efficacy of IIT-SIT to mitigate active dengue transmission. Specifically, the study will determine whether the release of male Wolbachia-infected Aedes aegypti mosquitoes can curtail the growth of dengue clusters, defined operationally by the Singapore National Environment Agency (NEA) as two or more reported dengue cases within a 150-meter radius and with illness onset dates within 14 days of each other. This study will randomize eligible clusters into intervention/control arms in real-time. Clusters assigned to the intervention arm will receive IIT-SIT treatment until cluster extinction (i.e. when no further cases are linked to the cluster). This trial closely mimics how IIT-SIT could be used as an additional tool for outbreak management, by treating areas with active dengue transmission in real-time. Conventional vector control measures will be carried out as per NEA's usual outbreak management practices in both intervention and control clusters. The intervention efficacy will be estimated through two primary endpoints: (1) probability of cluster extinction, as estimated from the time-to-cluster extinction among intervention versus control clusters; and (2) final size of the dengue cluster, as estimated by the difference in the final number of dengue cases in intervention versus control clusters.

This study will provide evidence from a randomized controlled trial for the efficacy of IIT-SIT in curbing ongoing transmission and provide an epidemiological basis for integrating IIT-SIT into the existing arsenal of outbreak management tools. The trial will assess the technology's feasibility for operationalization, and identify difficulties in implementation prior to larger-scale use for outbreak control.

ELIGIBILITY:
Eligible dengue clusters will be limited to public housing estates and with at least 10 dengue cases comprising that dengue cluster before allocation into intervention or control arms. The selected clusters will be in areas with relatively high sector-level GAI of at least 0.2 at the time of the 10th reported case. Additionally, the first 10 cases must be reported within 30 days of the first case. Additionally, clusters must be in areas which have never experienced Wolbachia-Aedes releases and at least 700 m away from existing Wolbachia-Aedes release areas.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2028-01-20 (Estimated)

PRIMARY OUTCOMES:
Impact of male Wolbachia-Aedes deployments on the time to cluster extinction | Up to 3 years
  In this analysis, male Wolbachia-Aedes exposure will be considered as a binary classification based on whether the dengue cluster is allocated to the intervention or control arm. Cox proportional hazards models will be used to assess the intervention effect of male Wolbachia-Aedes by estimating the hazards ratio, which compares the probability of cluster extinction between arms from following up clusters from enrolment to cluster extinction.
Impact of male Wolbachia-Aedes deployments on final cluster size, as measured by the difference in final cluster size between arms | Up to 3 years
  In this analysis, male Wolbachia-Aedes exposure will be considered as a binary classification based on whether the dengue cluster is allocated to the intervention or control arm. Negative binomial models will be used to assess the intervention effect of male Wolbachia-Aedes by estimating the average treatment effect of the intervention on the final number of dengue cases in intervention versus control clusters.

SECONDARY OUTCOMES:
Impact of male Wolbachia-Aedes deployments on the prevalence of Ae. aegypti/Ae. albopictus mosquitoes | Up to 3 years
  The study will test whether male Wolbachia-Aedes deployments will effectively suppress Ae. aegypti mosquito populations as well as whether they have an off-target impact on Ae. albopictus mosquito populations in intervention vs. control clusters.
Impact of male Wolbachia-Aedes deployments on dengue risk in clusters, measured by odds ratio of Wolbachia exposure distribution among laboratory-confirmed reported dengue cases compared to test-negative controls | Up to 3 years
  In this analysis, male Wolbachia-Aedes exposure will be considered as a binary classification based on whether a patient's residence is in an dengue cluster receiving intervention or a control cluster, where residence is defined as the primary place where the patient resided at reporting date.
Impact of male Wolbachia-Aedes deployments on the individual level reproduction number | Up to 3 years
  In this analysis, the researchers will use notified and individually geolocated dengue cases to calculate the spatially adjusted time-varying reproduction number, which estimates the number of forward infections caused by an individual.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ching Ng Group Director (Environmental Health Institute), PhD, Principal Investigator — Environmental Health Institute
Locations (1):
- National Environment Agency, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No